CLINICAL TRIAL: NCT02017249
Title: A Double-Blinded Randomized Placebo-Controlled Trial Exploring the Efficacy of Oral ARginine Supplementation to Improve Cellular Immune Function in Patients With Glioblastoma Multiforme
Brief Title: Efficacy Study of Oral Arginine to Improve Immune Function in Glioblastoma Multiforme
Acronym: ArginineGBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1364
Record Dates: First submitted 2013-11-07; First posted 2013-12-20 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2018-05

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Arginine; Silicon Dioxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arginine (Experimental): 24.15g of arginine supplement in powder form will be administered orally 3 times per day for 7 days before surgery and 7 days after surgery.
  Interventions: Drug: arginine in powder form
- Silica and cellulose placebo powder (Placebo Comparator): 3.5 teaspoons of placebo powder will be mixed with a sweet beverage and given orally 3 times per day for 7 days prior to surgery and 7 days after surgery.
  Interventions: Drug: Silica and cellulose placebo powder

INTERVENTIONS:
Drug: arginine in powder form
  Arms: Arginine
Drug: Silica and cellulose placebo powder
  Arms: Silica and cellulose placebo powder

SUMMARY:
The purpose of this study is to learn more about the ability of a substance called arginine to improve the functioning of the immune system in people with a certain type of brain tumor. This could lead to improvements in a type of treatment for brain tumors called immunotherapy. The immune system includes organs, cells, and substances in the body that fight infection and disease. Immunotherapy is a type of treatment that uses the immune system as a tool to seek out and destroy abnormal cells. Immunotherapy requires that the immune system be working properly. Arginine is a normal component of protein (an amino acid) that we all consume in foods such as red meat, poultry, fish, and dairy products and that our bodies can make. Arginine helps the immune system function normally. Recent research has shown that certain types of brain tumors decrease the amount of arginine in the body leading to impaired immune system function. This may interfere with the ability of immunotherapy to fight abnormal cells. We would like to see if giving people with brain tumors arginine in powder form will make their immune systems work better.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. Imaging consistent with GBM without clinical indication for primary CNS lymphoma or abscess, as determined by the treating physician.
3. Patient must be planned to proceed to definitive surgery intended for tumor resection, rather than needle biopsy, within a reasonable time frame from initial evaluation (7-14 days).
4. Patient must be neurologically stable, allowing for reasonable time frame between initial evaluation and subsequent surgical procedure (7-14 days).
5. Patient must have initial KPS greater than 80.
6. At the time of initial evaluation the patient must be on a stable dose of steroid medication if indicated.
7. Patient must have laboratory values, as determined by institutional controls, within the following parameters:

   * White blood cell count above lowest level for normal range
   * Renal function within normal limits (creatinine, BUN)
   * Liver function within normal limits (AST/ALT, total bilirubin, alkaline phosphatase)
8. Written informed consent is obtained prior to initiation of study procedures.

Exclusion Criteria:

1. Known autoimmune condition, underlying immune disease, or use of immunomodulatory prescription drugs (aside from steroids) for any medical condition.
2. Prescribed vasodilator medications: Phosphodiesterase Inhibitors: Sildenafil (Viagra), Nitrates, Alpha blockers: Terazosin (Hytrin), doxazosin (Cardura), alfuzosin (Uroxatral), tamsulosin (Flomax), and prazosin (Minipress).
3. Glaucoma
4. Known Herpes simplex virus (i.e. cold sores)
5. History of myocardial infarction or coronary artery disease.
6. Known allergy or intolerance to arginine.
7. Uncontrolled or poorly controlled seizures.
8. KPS less than 80.
9. Known renal or hepatic insufficiency or failure.
10. Known deficiency or dysfunction of intestinal absorption or motility.
11. History of other malignancy regardless of current status or treatment.
12. Underlying psychiatric condition or altered mental status that would violate stringent acquisition of informed consent or potentially preclude, in the opinion of the investigator, compliance with study requirements
13. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10-06 (Actual)

PRIMARY OUTCOMES:
Change in GBM patients immune function through arginine supplementation | study day 0 and 8
  25% increase in the functional response of peripheral T cells
Change in control group immune function through arginine supplementation | Study days 0 and 8
  Observe the change in T cell functional response

CONTACTS AND LOCATIONS:
Overall Officials: Allen Waziri, MD, Principal Investigator — Inova Health Care Systems
Locations (1):
- Inova Outpatient Surgery Clinic and Inova Fairfax Hospital, Fairfax, Virginia, United States